CLINICAL TRIAL: NCT06394245
Title: Determining the Effect of Progressive Relaxation Exercises on Postoperative Pain in Laparoscopic Living Kidney Donors
Brief Title: Progressive Relaxation Exercises for Kidney Donors
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fenerbahce University (Other)
Responsible Party: Principal Investigator, Ogr. Uyesi Naile, assit. prof., Fenerbahce University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2020 (2020/45)
Record Dates: First submitted 2024-04-25; First posted 2024-05-01 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Kidney Transplant; Complications; Muscle Relaxation

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): All sampled patients will administer STAI-1 and then VAS before relaxation exercises. Pain levels will be evaluated by applying VAS again. VAS and STAI will applie again to all patients at discharge. 400 mg contramol in 100 cc SF at 5cc/hour continues on the first day after surgery by PCA (Patient control analgezia). The total number of boluse administrations and additional analgesic requirements of the patients will record by PCA after the application during the day. After the implementation of the PMR exercise protocol, no side effects or signs of discomfort will observe in the patients. In the hospital where the study will conduct, if patients can tolerate it, they are routinely mobilized for 8 hours after surgery and are fed there 6 hours later. Patients in the experimental and control groups will evaluate in terms of postoperative mobilization and oral feeding initiation times.
  Interventions: Other: Progressive muscle exercises
- Control Group (No Intervention): Patients in the control group will not receive any special intervention, only routine care. After data will collect from the patients in the control group, they will be informed that they can do progressive muscle relaxation exercises whenever they want.

INTERVENTIONS:
Other: Progressive muscle exercises — The initiative was made with the Turkish Psychologists Association's Progressive Relaxation Exercises audio recorded. PGE consists of a recording of breathing exercises and progressive muscle stretching exercises, with music in the background that will relax the patient. The first part of the recordings takes approximately 10 minutes. It continues and includes information about the definition of relaxation exercise, its purpose, benefits and points to consider when starting the exercises, correct breathing in the appropriate position and what the environment should be like. The second part consists of how to contract and relax certain muscles in our body, which takes approximately 25-30 minutes, and the steps to exit this process after the relaxation session is over.
  Arms: Experimental group

SUMMARY:
Complex emotions and other possible changes associated with agreeing to enroll after laparoscopic donor nephrectomy may cause living donors to experience anxiety, increase in perceived pain temperature, or last longer after surgery.

Purpose: The purpose of using this method is to determine the effect of progressive relaxation exercises on postoperative pain in laparoscopic living kidney donors.

Method: This randomized controlled single-blind study will conduct with 63 patients (study group = 31, control group = 32) who met the care inclusion criteria and underwent laparoscopic living donor nephrectomy in the transplantation service of a private hospital in Istanbul. The sample size and power of the study were calculated with power analysis (G*Power 3.1). The data will obtain in the study will evaluate in a computer environment through the SPSS 22.0 statistical program. The data of the research will combine with the patient information formula, postoperative patient follow-up and evaluation formula, Visual Pain Scale (VAS), PCA and total demand and delivery of boluses and additional analgesic procedures. This study was conducted in accordance with CONSORT.

DETAILED DESCRIPTION:
According to 2021 data, 62% of kidney transplants in the world are performed from cadavers. In Turkey, due to the low number of cadaver organ donations, living kidney transplants are more common (91.17%). Although laparoscopic donor nephrectomy is a minimally invasive technique that offers less pain, better cosmetic results and lower morbidity rates worldwide, living kidney donors experience postoperative pain that hinders postoperative recovery and creates anxiety and fear in some. Lack of direct benefit to the individual, fear of losing the healthy kidney and death after surgery, complex feelings about accepting the transplant, and other possible complications may cause living donors to experience post-operative anxiety, increased perceived pain intensity, or prolonged duration. Furthermore, although acute postoperative pain is an expected outcome after most elective surgeries, including donor nephrectomy, it has been recognized that inadequately treated postoperative acute pain can develop into chronic pain, which is often misdiagnosed and neglected. While this rate was 5.7% after laparoscopic living donor nephrectomy in the study by In one study it was 41% in the study . These conditions may negatively affect the return to normal life and the patients' quality of life. This pain in donors is tried to be managed with opioid and non-opioid medications, social support and ambulation. These efforts have proven challenging, as the subjective nature of pain perception further complicates the ability to achieve satisfactory pain control. Additionally, studies have indicated that certain patient comorbidities and social factors may cause an increase in patients' pain perception.Progressive relaxation exercise (PGE) is a type of exercise that provides tension and relaxation of a large muscle group, developed 1920. In the literature, it is stated that PGE application makes it easier for the individual to cope with pain due to reasons such as reducing muscle tension, anxiety and stress effects, reducing blood pressure, heart rate, lactic acid production, increasing concentration and positive thoughts by regulating the activity of the nervous system, suppressing negative thoughts, and diverting attention. stated. When we look at the literature, there are almost no studies discussing non-pharmacological methods to prevent or reduce pain in donors, which is thought to be mostly psychosomatic. RCTs using standardized relaxation protocols are needed to provide further evidence on this topic. In the light of this information, the aim of this study is to determine the effect of progressive relaxation exercises on postoperative pain in laparoscopic living kidney donors.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study Literate and knowing the native language

Exclusion Criteria:

* Chronic pain history Patients who developed complications during surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2024-05-15 (Estimated); Primary Completion 2024-05-25 (Estimated); Study Completion 2024-06-15 (Estimated)

PRIMARY OUTCOMES:
Hypothesis | Two days
  Performing progressive relaxation exercises after donor nephrectomy will reduce the postoperative VAS pain score in patients.

REFERENCES:
- [Derived] Akinci N. Effect of progressive muscle relaxation on postoperative pain in laparoscopic living kidney donors: a randomized controlled trial. BMC Surg. 2025 Sep 24;25(1):410. doi: 10.1186/s12893-025-03187-y. PMID 40993691